CLINICAL TRIAL: NCT01109836
Title: ASPIS-Austrian Polyintervention Study to Prevent Cognitive Decline After Ischemic Stroke
Brief Title: Austrian Polyintervention Study to Prevent Cognitive Decline After Ischemic Stroke
Acronym: ASPIS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Danube University Krems (Other)
Collaborators: NÖ Forschungs- und Bildungsges.m.b.H (NFB) (Unknown)
Responsible Party: Prim. Univ. Prof. Dr. Michael Brainin, Danube University Krems
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: DUK-2010-001; LS 09-002 (Other Grant/Funding Number: Life Science Krems)
Record Dates: First submitted 2010-04-15; First posted 2010-04-23 (Estimated); Last update posted 2015-01-13 (Estimated); Status verified 2010-06

CONDITIONS: Ischemic Stroke; Cognitive Decline; Dementia
Keywords: prevention; cognitive decline; post-stroke dementia; life-style intervention; vascular risk factors; polyintervention; multifactorial treatment
MeSH Terms: conditions — Ischemic Stroke; Cognitive Dysfunction; Dementia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Motivation and lifestyle intervention (Experimental): Intensive control and motivation for better compliance with medication, regular blood pressure measurements, diet changes and physical activity.
  Interventions: Behavioral: Motivation and lifestyle intervention
- Control (No Intervention): Standard stroke care

INTERVENTIONS:
Behavioral: Motivation and lifestyle intervention — Intensive control and motivation for better compliance with medication, regular blood pressure measurements, diet changes and physical activity.
  Arms: Motivation and lifestyle intervention

SUMMARY:
Aim of this randomized controlled study is to test if intensive polyintervention therapy including life style modifications targeting at reduction of modifiable risk factors of stroke can reduce the risk of post-stroke cognitive decline compared to a group of patients receiving standard care.

DETAILED DESCRIPTION:
Stroke is the second most frequent cause of death and cognitive deficits including dementia occur frequently following a stroke. The frequency of cognitive disturbances has been reported up to 30% and thus occurs three times more frequent than recurrent stroke (10%). Major attempts have been made to prevent the occurrence of new strokes by means of effective strategies including preventive drugs. In contrast, hardly any studies have been performed addressing the prevention of deteriorating cognitive function following a stroke. In spite of this high prevalence therapeutic possibilities are extremely limited. It must be expected that cognitive deficits become even a more frequent disability following stroke. This is caused by the increased aging of the population leading to further increase of incidence, furthermore that more people survive their acute stroke due to increased possibilities of acute treatment, and that frequent risk factors (e.g. hypertension, diabetes) are increasingly controlled, thus leading to less severe strokes with less severe and permanent motor deficits, but an increase of potentially disabling cognitive disturbances. The aim of this randomized controlled study is to test an intensive multiple intervention therapy for the first time in stroke and to add life style modifications targeting modifiable risk factors for cognitive deterioration.

It is hypothesized that the risk of post-stroke cognitive decline can be significantly reduced compared to a control group with standard care when using polyintervention. These interventions will focus on nutrition, exercise, cognitive and social activity and monitoring and management of metabolic and vascular risk factors. Regular contacts with the subjects shall increase motivation and adherence to the study protocol.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic ischemic stroke with clinical syndrome of stroke and a corresponding ischemic lesion.
* MRI or CT results compatible with clinical diagnosis of acute ischemic stroke
* NIH Stroke Scale Score on admission 1 to 14, both inclusive
* Modified Rankin Scale before stroke 0 to 2, inclusive
* Randomization within 3 months after stroke onset (goal: 80% within 3 weeks)
* Sufficient communication possible
* Informed consent given by the patient and/or the patient's legally acceptable representative

Exclusion Criteria:

* Substantial cognitive decline (Mini Mental State Examination (MMSE) score > 24) or pre-existing dementia or Parkinson disease
* Persistent disturbed level of consciousness
* Persistent aphasia
* Pre-existing significant psychiatric diseases (i.e. Schizophrenia, Major Depression, Bipolar Disorders, all according to DSMIV); Patients with minor Depression (DSM IV) can be included
* Severe sensory impairment making neuropsychological testing impossible
* Severe comorbidity (e.g. unstable or severe cardiovascular or pulmonal disease, neoplasm, severe liver or renal insufficiency and symptomatic stenosis of the ipsilateral carotid artery, cancer…)
* Unreliability for follow up
* Unwillingness or inability to participate or to sign the informed consent

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2010-06; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Number of persons having cognitively declined at 24 months | 24 months after randomization
  Cognitive decline is defined as a significant decline in the composite scores of at least 2 of 5 neuropsychologically tested domains (speed of mental processing, executive functions, working memory, memory, spatial constructive functions). The alpha level for the decision is 0.05.
Cognitive decline measured on the Cognitive Subscale of the Alzheimer's disease assessment scale (ADAS-cog) at 24 months | 24 months after randomization
  Difference between the measures at baseline and at 24 months on the Cognitive Subscale of the Alzheimer's disease assessment scale (ADAS-cog).

SECONDARY OUTCOMES:
Number of persons having cognitively declined 12 months after randomization | 12 months after randomization
  Cognitive decline is defined as a significant decline in the composite scores of at least 2 of 5 neuropsychologically tested domains (speed of mental processing, executive functions, working memory, memory, spatial constructive functions). The alpha level for the decision is 0.05.
Cognitive decline on the Cognitive Subscale of the Alzheimer's disease assessment scale (ADAS-cog) at 12 months | 12 months after randomization
  Difference between the measures at baseline and at 12 months on the Cognitive Subscale of the Alzheimer's disease assessment scale (ADAS-cog).
Cognitive impairment on the Mini-Mental-State-Examination (MMSE) scale at 12 months | 12 months after randomization
Cognitive impairment on the Mini-Mental-State-Examination (MMSE) scale at 24 months | 24 months after randomization
Change in cognitive abilities measured by composite scores for each of 5 cognitive domains | 12 months after randomization
  For each of the five cognitive domains (executive functions, working memory, general memory, speed of cognitive processing, visual spatial ability) standardized composite scores are calculated from the differences between baseline and 12 months in individual neuropsychological test results.
Composite outcome for vascular events | 24 months after randomization
  vascular events include recurrent stroke, ACS, bypass surgery, PTA and vascular death
Neurological status on the National Institute of Health Stroke Scale (NIHSS) score | 12 months after randomization
Functional status on the modified Rankin Scale | 12 months after randomization
Activities of daily living on Barthel Index | 12 months after randomization
Quality of life on the EQ-5D | 12 months after randomization
Depression on the Center for Epidemiologic Studies Depression Scale (CESD) | 12 months after randomization
All cause mortality | 24 months after randomization
Change in cognitive abilities measured by composite scores for each of 5 cognitive domains | 24 months after randomization
  For each of the five cognitive domains (executive functions, working memory, general memory, speed of cognitive processing, visual spatial ability) standardized composite scores are calculated from the differences between baseline and 24 months in individual neuropsychological test results.
Neurological status on the National Institute of Health Stroke Scale (NIHSS)score | 24 months after randomization
Functional status on the modified Rankin Scale | 24 months after randomization
Activities of daily living on Barthel Index | 24 months after randomization
Quality of life on the EQ-5D | 24 months after randomization
Depression on the Center for Epidemiologic Studies Depression Scale (CESD) | 24 months after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Michael Brainin, Prof. MD, Principal Investigator — Danube University Krems
Locations (5):
- Austria (5):
  - Dept of Neurology Landesklinikum Waldviertel Horn / Allentsteig, Horn
  - Dept of Neurology, Landesklinikum Mostviertel Amstetten-Mauer, Mauer bei Amstetten
  - Dept. Neurology, LK St.Pölten, Sankt Pölten
  - Dept of Neurology, Landesklinikum Donauregion Tulln, Tulln
  - Dept of Neurology, Landesklinikum Wr. Neustadt, Wiener Neustadt

REFERENCES:
- [Derived] Matz K, Tuomilehto J, Teuschl Y, Dachenhausen A, Brainin M. Comparison of oral glucose tolerance test and HbA1c in detection of disorders of glucose metabolism in patients with acute stroke. Cardiovasc Diabetol. 2020 Dec 5;19(1):204. doi: 10.1186/s12933-020-01182-6. PMID 33278898
- [Derived] Matz K, Teuschl Y, Firlinger B, Dachenhausen A, Keindl M, Seyfang L, Tuomilehto J, Brainin M; ASPIS Study Group. Multidomain Lifestyle Interventions for the Prevention of Cognitive Decline After Ischemic Stroke: Randomized Trial. Stroke. 2015 Oct;46(10):2874-80. doi: 10.1161/STROKEAHA.115.009992. Epub 2015 Sep 15. PMID 26374482
- [Derived] Brainin M, Matz K, Nemec M, Teuschl Y, Dachenhausen A, Asenbaum-Nan S, Bancher C, Kepplinger B, Oberndorfer S, Pinter M, Schnider P, Tuomilehto J; ASPIS Study Group. Prevention of poststroke cognitive decline: ASPIS--a multicenter, randomized, observer-blind, parallel group clinical trial to evaluate multiple lifestyle interventions--study design and baseline characteristics. Int J Stroke. 2015 Jun;10(4):627-35. doi: 10.1111/ijs.12188. Epub 2013 Nov 10. PMID 24206541